CLINICAL TRIAL: NCT03458091
Title: Evaluation of Lung Atelectasis During Apneic Oxygenation Using Trans Nasal Humidified Rapid Insufflation Ventilatory Exchange (THRIVE) in Adults During Laryngeal Surgery.
Brief Title: Evaluation of Lung Atelectasis During Apneic Oxygenation Using THRIVE in Adults During Laryngeal Surgery.
Acronym: A-THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, Senior Consultant, Associate Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-THRIVE
Record Dates: First submitted 2018-01-21; First posted 2018-03-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Tobacco Use Cessation Devices; Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubation (Active Comparator): The patients will be intubated and ventilated
  Interventions: Device: Endotracheal intubation
- THRIVE (Experimental): The patients will be oxygenated during apnea using THRIVE
  Interventions: Device: THRIVE

INTERVENTIONS:
Device: THRIVE — Oxygenation during apnea using transversal humidified oxygen
  Arms: THRIVE
Device: Endotracheal intubation — Ventilation during the procedure is governed by an endotracheal tube in the trachea and mechanical ventilation
  Arms: Intubation

SUMMARY:
Oxygenation with high-flow nasal cannula with 100% oxygen have now been evaluated in a number of studies and the data are convincing. The THRIVE technique is able to oxygenate patients safely and vital parameters has been shown to be stable. But it is of great importance to evaluate this new concept regarding other potential negative physiological aspects such as lung atelectasis and inflammatory stress response before implementing it into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, >18 years old.
2. ENT-surgery where apnea is of benefit for the surgeon (eg. intraoral or laryngeal surgery).
3. Capable of understanding the study information and sign the written consent.

Exclusion Criteria:

1. ASA>2
2. NYHA >2
3. Pacemaker or ICD.
4. BMI >35
5. Pregnancy
6. Manifest cardiac failure or coronary disease
7. Severe gastrointestinal reflux.
8. Neuromuscular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Electrical impedans tomography | baseline, intraoperative, 2 hours after start of intervention
  Changes in lung volumes

SECONDARY OUTCOMES:
Difference in Endtidal and arterial carbon dioxide partial pressure in the end of the procedure | max 30 minutes after start of intervention
  Difference in Endtidal and arterial carbon dioxide partial pressure in the end of the procedure
Increase in arterial carbon dioxide during the apnea | max 30 minutes after start of intervention
  Measurement of arterial blood gases and here arterial carbon dioxide

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided